CLINICAL TRIAL: NCT07133594
Title: Validation of a French-language Questionnaire for Patient Experience in Radiotherapy
Brief Title: Validation of a Questionnaire in the French Language for the Patient Experience in Radiotherapy
Acronym: QF-EXPERT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET24-354 - QF-EXPERT; 2024-A02830-47 (Other: ID-RCB)
Record Dates: First submitted 2025-07-31; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Validation RTEQ (RadioTherapy Experience Questionnaire) in French; Patients Requiring Radiotherapy
Keywords: RTEQ; Questionnaire validation; French translation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Questionnaires for patients receiving 10 or fewer radiotherapy sessions_ (Experimental): Patients receiving 10 or fewer radiotherapy sessions: Patient will complete two questionnaires only once between Day 2 and Day 7.
  Interventions: Other: RTEQ (RadioTherapy Experience Questionnaire) in French; Other: EORTC PATSAT-C33 questionnaire
- Questionnaires for patients receiving 11 or more radiotherapy sessions_ (Experimental): Patients receiving 11 or more radiotherapy sessions. They will complete two questionnaires, at two measurement times: between Day 2 and Day 7 and then during the last week.
  Interventions: Other: RTEQ (RadioTherapy Experience Questionnaire) in French; Other: EORTC PATSAT-C33 questionnaire

INTERVENTIONS:
Other: RTEQ (RadioTherapy Experience Questionnaire) in French — Complete the RTEQ questionnaire translated and adapted to the French language in patients receiving external radiotherapy. Depending on the number of radiotherapy sessions received, the questionnaire will be completed 1 or 2 times during the study.
Other: EORTC PATSAT-C33 questionnaire — Complete the EORTC-PATSAT-C33 questionnaire after completing the RTEQ questionnaire. Depending on the number of radiotherapy sessions received, the questionnaire will be completed 1 or 2 times during the study.

SUMMARY:
More than 50% of cancer patients have radiotherapy (RT) as part of their care pathway. Scientific and technological advances leads to an increase in demand. The development of hypofractionation is also increasing the capacity to treat more patients. These transformations raise questions from an organizational point of view, the quality of care and the response to patient needs.

Several publications highlight that evaluating patient's experience, satisfaction, and collecting their ideas are excellent foundations for delivering patient-centered care (3,4). To assess the patient experience in RT, Olausson et al. developed and validated a questionnaire in English. To this day , this questionnaire has not been validated in French.

The main objective is to validate the psychometric property of reliability of the Radiotherapy Experience Questionnaire (RTEQ) after its adaptation into French. This project also includes an assessment of patient satisfaction regarding their RT care pathway.

This study is part of a broader initiative aimed at redesigning the patient journey in radiotherapy, and innovating in the tools and in the overall care approach.

DETAILED DESCRIPTION:
There will be 4 steps in this study.

* Phase 1: the RTEQ has been adapted into French by a working group. Phase alreaday completed.
* Phase 2: this is the RTEQ pre-test translated into French. Currently in progress. Comprehension of the questionnaire will be assessed in 50 patients at the Centre Leon Berard (CLB) to obtain the final French version. Patients will complete the RTEQ and a debriefing questionnaire at a time. Patients undergoing hypofractionated RT (between 2 and 10 sessions) as well as patients with more than 11 sessions will be included. Patients undergoing hypofractionated RT will complete the questionnaire at the penultimate session. Patients with at least 11 sessions will be included and will complete the questionnaire during the last week of treatment. The debriefing questionnaire has been developed to determine whether the questionnaire is too long, whether each questions are clear and comprehensive or not.
* Phase 3: pre-test analysis. A descriptive analysis of the responses to each item, as well as the debriefing questionnaire, will be carried out. A meeting with the working group will decide on the necessary modifications for a final version.
* Phase 4: Paucicentric study + validation of the psychometric properties of the RTEQ in French.

Patients will complete the RTEQ and the EORTC PATSAT-C33 questionnaire.

* Group 1: For patients undergoing hypofractionated RT: one measurement period, between Days 2 and 7 (Time n°1).
* Group 2: For patients with at least 11 sessions, two measurement periods: during the first week between Days 2 and 7 (Time n°1) and then during the last week (Time n°2).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Patient requiring curative external radiotherapy (at least 2 sessions)
* Patient covered by a medical insurance
* Patient informed and not opposing to the study

Exclusion Criteria:

* Patient who don't understand or can't read French
* Any congitive impairment or condition likely to limit the use of scales and questionnaires
* Patient requiring tutorship or curatorship or patient deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To validate the psychometric reliability property (internal consistency between items) of the RTEQ questionnaire after translation and adaptation to the French language for the evaluation of the experience of patients receiving external RT. | Time n°1 : Between Day 2 and Day 7 of radiotherapy
  Cronbach's alpha coefficient for each dimension of the RTEQ from the questionnaire items at Time n°1 (T1)

SECONDARY OUTCOMES:
Other psychometric properties of the questionnaire | Time n°1 : between Day 2 and Day7 of radiotherapy for all patients; Time n°2 : during the last week of radiotherapy if patient have more than 10 sessions of radiotherapy
  The validity of the content of the questionnaire (associated criterion: distribution of RTEQ items at Time n°1); The structural validity of the questionnaire (associated criterion: items of the RTEQ questionnaire at Time n°1, confirmatory factor analysis); Comparison of known groups: comparison between patients with hypofractionated RT: maximum 10 sessions (group 1) versus those with more than 10 sessions (group 2) (associated criterion: scores of each RTEQ scale at Time n°1 for group 1 vs Time n°2 for group 2); Convergent and divergent validity (associated criterion: correlation matrix between RTEQ scores vs satisfaction scores of the EORTC PATSAT-C33 questionnaire)
The level of satisfaction of patients treated by RT from the EORTC PATSAT-C33 questionnaire | Time n°1: between Day 2 and Day 7 of radiotherapy
  Scores of each scale of the PATSAT-C33 at Time n°1 (scale graduated from 1 to 5)
The evolution of satisfaction between the first and last week of treatment for patients in group 2 | Time n°1: between Day 2 and Day 7 of radiotherapy for all patients; Time n°2: during the last week of radiotherapy if patient receive more than 10 sessions of radiotherapy
  PATSAT-C33 scores at Time n°1 and Time n°2
The impact of the number of RT sessions on the measurement of satisfaction: comparison between patients in group 1 versus those in group 2 | Time n°1: between Day 2 and Day 7 of radiotherapy for all patients; Time n°2: during the last week of radiotherapy if patient receive more than 10 sessions of radiotherapy
  Scores of each scale of the PATSAT-C33 at Time n°1 for group 1 vs Time n°2 for group 2

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BOISBOUVIER, Msc R&I in Healthcare (RT), Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Leon Berard, Lyon, France

IPD SHARING:
Plan to Share IPD: No